CLINICAL TRIAL: NCT03502889
Title: Single Dose Adductor Canal Block With SPANK (Sensory Posterior Articular Nerves of the Knee) Block Compared to Single Dose Adductor Canal Block and Pain Control After Total Knee Arthroplasty
Brief Title: Single Dose Adductor Canal Block vs SPANK Block for TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Angela Curell, Anesthesiology Resident, San Antonio Uniformed Services Health Education Consortium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPANK Block
Record Dates: First submitted 2018-03-13; First posted 2018-04-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Osteo Arthritis Knee; Pain, Postoperative; Pain, Acute
Keywords: Total Knee Arthroplasty; SPANK Block; Adductor Canal Block; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block Alone (Active Comparator): Control arm to receive Adductor Canal Block without additional interventions Intervention: ropivacaine 0.5% 15cc injected under ultrasound guidance
  Interventions: Procedure: Adductor Canal Block; Drug: Ropivacaine Hcl 0.5% Inj Vil 30Ml; Device: Pajunk sonoplex stim needle
- SPANK Block Plus Adductor Canal Block (Experimental): Experimental arm to receive Adductor Canal Block plus SPANK Block (Sensory Posterior Articular Nerves of the Knee) without additional interventions Intervention: ropivacaine 0.5% 15cc injected under ultrasound guidance into the adductor canal plus 20cc ropivacaine 0.5% injected into the posterior tissues of the knee
  Interventions: Procedure: SPANK Block (Sensory Posterior Articular Nerves of the Knee); Procedure: Adductor Canal Block; Drug: Ropivacaine Hcl 0.5% Inj Vil 30Ml; Device: Pajunk sonoplex stim needle

INTERVENTIONS:
Procedure: SPANK Block (Sensory Posterior Articular Nerves of the Knee) — Injection of local anesthetic into the tissues on the posterior aspect of the knee to provide sensory blockade of the articular nerves of the knee.
  Arms: SPANK Block Plus Adductor Canal Block
Procedure: Adductor Canal Block — Injection of local anesthetic into the inner thigh under ultrasound guidance to provide sensory blockade to the anterior aspect of the knee
Drug: Ropivacaine Hcl 0.5% Inj Vil 30Ml — Amide local anesthetic, this concentration is commonly used to achieve surgical level anesthesia. The drug itself is not being studied and the same concentration will be used in all participants.
Device: Pajunk sonoplex stim needle — Echogenic needle used for ultrasound guided nerve blockade.

SUMMARY:
This is a prospective, randomized control trial to compare SPANK block combined with adductor canal block to adductor canal block alone in treatment of post-operative pain after total knee arthroplasty. The primary outcome is pain control, which will be measured throughout the post-operative course using morphine equivalents of opioid analgesics used during the first 24 hours after surgery. Secondary outcomes include pain scores recorded at 4, 8, 12, 16, 20, and 24 hours post-operatively, cumulative pain score, incidence of post-operative nausea and vomiting, and extent of motor blockade. The study will aid in answering the question of whether SPANK block is an effective adjunct in preventing pain and decreasing opioid requirement after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40 and 80 years old undergoing total knee arthroplasty amenable to peripheral nerve block for perioperative analgesia.
* BMI <45
* ASA class III or less

Exclusion Criteria:

* Inability to sign consent form
* Allergy to medications used in the study
* Repeat surgery
* History of seizure disorder
* Simultaneous bilateral TKA
* History of substance abuse
* BMI >45
* Opioid consumption of greater or equal to 30mg morphine equivalents per day
* Age <40 or >80 years old
* ASA IV or greater
* Inability to use a PCA
* Inability to access the intrathecal space
* Infection at the site of injection (either for spinal or PNB)
* INR greater than or equal to 1.4

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Opioid Consumption | 24 hours postoperatively
  Amount of opioids used within the first 24 hours post-operatively, starting from when the patient leaves the operating room, measured in PO morphine equivalents

SECONDARY OUTCOMES:
Postoperative Pain Scores | 4, 8, 12, 16, and 24 hours postoperatively
  Verbal pain score measured via numerical rating scale from 1-10 at 4 hrs, 8 hrs, 12hrs, 16hrs, and 24 hours.
Time to first opioid use | 24 hours postoperatively
  The amount of time measured from when the patient leaves the operating room to the time when they receive their first dose of any opioid medication.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Curell, MD, Principal Investigator — San Antonio Uniformed Services Health Education Consortium

IPD SHARING:
Plan to Share IPD: Undecided
If shared, will plan to provide. All IPD that underlie results in publication
  * Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form (ICF)
  * Clinical Study Report (CSR)
  Starting 6 months after publication

REFERENCES:
- [Background] Terkawi AS, Mavridis D, Sessler DI, Nunemaker MS, Doais KS, Terkawi RS, Terkawi YS, Petropoulou M, Nemergut EC. Pain Management Modalities after Total Knee Arthroplasty: A Network Meta-analysis of 170 Randomized Controlled Trials. Anesthesiology. 2017 May;126(5):923-937. doi: 10.1097/ALN.0000000000001607. PMID 28288050
- [Background] Gao F, Ma J, Sun W, Guo W, Li Z, Wang W. Adductor Canal Block Versus Femoral Nerve Block for Analgesia After Total Knee Arthroplasty: A Systematic Review and Meta-analysis. Clin J Pain. 2017 Apr;33(4):356-368. doi: 10.1097/AJP.0000000000000402. PMID 27322397
- [Background] Wang D, Yang Y, Li Q, Tang SL, Zeng WN, Xu J, Xie TH, Pei FX, Yang L, Li LL, Zhou ZK. Adductor canal block versus femoral nerve block for total knee arthroplasty: a meta-analysis of randomized controlled trials. Sci Rep. 2017 Jan 12;7:40721. doi: 10.1038/srep40721. PMID 28079176
- [Background] Karlsen AP, Wetterslev M, Hansen SE, Hansen MS, Mathiesen O, Dahl JB. Postoperative pain treatment after total knee arthroplasty: A systematic review. PLoS One. 2017 Mar 8;12(3):e0173107. doi: 10.1371/journal.pone.0173107. eCollection 2017. PMID 28273133
- [Background] Li D, Ma GG. Analgesic efficacy and quadriceps strength of adductor canal block versus femoral nerve block following total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2016 Aug;24(8):2614-9. doi: 10.1007/s00167-015-3874-3. Epub 2015 Nov 26. PMID 26611901
- [Background] Bauer MC, Pogatzki-Zahn EM, Zahn PK. Regional analgesia techniques for total knee replacement. Curr Opin Anaesthesiol. 2014 Oct;27(5):501-6. doi: 10.1097/ACO.0000000000000115. PMID 25111605
- [Background] Pelt CE, Anderson AW, Anderson MB, Van Dine C, Peters CL. Postoperative falls after total knee arthroplasty in patients with a femoral nerve catheter: can we reduce the incidence? J Arthroplasty. 2014 Jun;29(6):1154-7. doi: 10.1016/j.arth.2014.01.006. Epub 2014 Jan 16. PMID 24581899
- [Background] Baratta JL, Gandhi K, Viscusi ER. Perioperative pain management for total knee arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):22-36. doi: 10.3113/jsoa.2014.0022. PMID 24641894
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Wasserstein D, Farlinger C, Brull R, Mahomed N, Gandhi R. Advanced age, obesity and continuous femoral nerve blockade are independent risk factors for inpatient falls after primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1121-4. doi: 10.1016/j.arth.2012.08.018. Epub 2012 Dec 21. PMID 23265274
- [Background] Feibel RJ, Dervin GF, Kim PR, Beaule PE. Major complications associated with femoral nerve catheters for knee arthroplasty: a word of caution. J Arthroplasty. 2009 Sep;24(6 Suppl):132-7. doi: 10.1016/j.arth.2009.04.008. Epub 2009 Jun 24. PMID 19553071